CLINICAL TRIAL: NCT06173206
Title: Effect of Single-course Malaria Chemoprevention on Clearance of and Protection from Plasmodium Falciparum Infection in the Presence of Resistance-associated Genotypes in Cameroon
Brief Title: Parasite Clearance and Protection from Infection (PCPI) in Cameroon
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2022-KEP-814
Record Dates: First submitted 2023-12-07; First posted 2023-12-15 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2024-06

CONDITIONS: Malaria
Keywords: Malaria; Perennial malaria chemoprevention (PMC); Intermittent preventative treatment of malaria in infants (IPTi); Sulfadoxine-pyrimethamine (SP); Chemoprevention; Drug resistance
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Intervention Model Description: Groups 1-2 will receive a 7-day course of placebo artesunate; Group 3 will be given a 7-day course of active artesunate. This will span Day -7, -6, -5, -4, -3, -2, and -1. Then, on Day 0, children in Groups 1-2 will receive a single course of malaria chemoprevention, whereas Group 3, having completed a 7-day course of AS will receive placebo SP.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Fully placebo controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Sulfadoxine-pyrimethamine (SP) (Active Comparator): Groups in the SP group will receive a 7-day course of placebo artesunate (at day -7, -6, -5, -4, -3, -2, and -1), followed by a single course of SP plus placebo AQ for 3 days.
  Interventions: Drug: SP (Macleods Pharmaceuticals Ltd)
- Sulfadoxine-pyrimethamine plus amodiaquine (SPAQ) (Active Comparator): Groups in the SPAQ group will receive a 7-day course of placebo artesunate (at day -7, -6, -5, -4, -3, -2, and -1), followed a single course of placebo SP placebo plus AQ for 3 days.
  Interventions: Drug: SPAQ (Guilin Pharmaceuticals)
- Artesunate monotherapy (AS) (Active Comparator): Groups in the AS group will receive a 7-day course of active artesunate (at day -7, -6, -5, -4, -3, -2, and -1), followed a single course of placebo SP plus placebo AQ for 3 days.
  Interventions: Drug: AS (Guilin Pharmaceuticals)

INTERVENTIONS:
Drug: SP (Macleods Pharmaceuticals Ltd) — Children who weigh <10kg will receive Sulfadoxine-pyrimethamine paediatric formulation (250mg/12.5mg) dispersable tablets; children who weigh >10kg will receive 500mg sulfadoxine plus 25mg pyrimethamine
  Arms: Sulfadoxine-pyrimethamine (SP)
Drug: SPAQ (Guilin Pharmaceuticals) — Children will receive 500mg sulfadoxine plus 25mg pyrimethamine as one tablet, and 153mg amodiaquine (as hydrochloride) as one tablet on Day 0, and Children will 153mg amodiaquine (as hydrochloride) as one tablet on days 1 and 2.
  Arms: Sulfadoxine-pyrimethamine plus amodiaquine (SPAQ)
Drug: AS (Guilin Pharmaceuticals) — Children will receive 4 mg/kg/day for 7 days
  Arms: Artesunate monotherapy (AS)

SUMMARY:
The Cameroon PCPI study will measure the effect of the parasite genotypes associated with SP resistance on parasite clearance and protection from infection when exposed to SP. The total number of participants is expected to be 900 healthy between 3 to 5 years old who have no symptoms of malaria infection of which 450 children will be assigned to the SP group, 250 to the SPAQ group, and 200 to the AS group. The results of this study will allow to measure the effect of the parasite genotypes associated with SP resistance on parasite clearance and protection from infection when exposed to SP.

DETAILED DESCRIPTION:
The World Health Organization (WHO) recently published new malaria chemoprevention guidelines that included a recommendation for the provision of perennial malaria chemoprevention (PMC) with sulfadoxine-pyrimethamine (SP) to children resident in areas of high malaria transmission. PMC is the successor to an intervention originally known to as intermittent preventive treatment of malaria in infants (IPTi) that involved SP dosing of children at 2, 3 and 9 months of age during vaccination visits of the Essential Programme on Immunization (EPI) that coincide with the 2nd and 3rd doses of the DPT/Penta and measles vaccines. Under the new PMC guidelines, countries are now encouraged to increase the number and frequency of SP doses, and to extend the target age beyond the first year of life.1 Evidence supporting PMC comes in part from meta-analysis2 of six randomised placebo-controlled trials3-8 that demonstrated the protective effect of SP against clinical malaria, anaemia, hospital admissions due to malaria infection, and all-cause hospital admissions. Biomarkers of SP resistance, however, vary in different malaria-endemic settings and have been shown to compromise its protective effect.

In East and Southern Africa, Plasmodium falciparum parasites carry a high frequency of mutations in the Pfdhfr and Pfdhps genes with differing degrees of effect. In Mozambique, for example, SP was protective against malaria infection despite the Pfdhps A437G plus K540E double mutation circulating in over one-half, 52.3%, of P. falciparum (Pf) parasites. 5,9,10 In contrast, SP showed no protective effect in an IPTi trial in Northeastern Tanzania11 where 94.3% of Pf parasites had Pfdhps K540E. However, in this trial, the Pfdhps A581G mutation was also present in 55.0% of Pf parasites, forming the haplotype ISGEGA at codons 431, 436, 437, 540, 581 and 613.12 Thus, Pf appears to be highly resistant to SP where the A581G mutation is concurrently expressed with K540E. Fortunately, for PMC with SP there are few locations in East Africa where the combination of K540E and A581G circulate; most areas across Central, East and Southern Africa have parasites that contain the K540E without the A581G mutation (Pfdhps haplotype ISGEAA). The prevalence threshold of the ISGEAA haplotype at which SP is no longer protective is unknown. Indeed, there may not be an upper limit, although empirical studies are needed to confirm this.

In West Africa, specifically the Sahel region, there are emerging parasite genotypes that harbour a distinct haplotype of Pfdhps, VAGKGS,13,14 which lacks the K540E. These observations have come from molecular monitoring conducted alongside the delivery of intermittent preventive treatment of malaria in pregnancy (IPTp) with SP, and seasonal malaria chemoprevention (SMC) that targets children under 5 years of age with a combination of SP plus amodiaquine (AQ). The VAGKGS haplotype, and the related VAGKAS and VAGKAA, have been reported in 2-40% of Pf parasites in Cameroon, Chad, Niger and Nigeria. The current distribution of parasites harbouring these genotypes is only partially described, and the effect these mutations have on parasite susceptibility to SP remains unknown. Nevertheless, it is possible that parasites harbouring Pfdhps-VAGKGS pose a threat to the effectiveness of PMC with SP or other SP-containing chemoprevention strategies in some parts of the West African Sahel. Thus, there are two clear evidence gaps, one in East/Southern Africa and another in West Africa, which the PCPI (parasite clearance and protection from infection) protocol has been developed to fill. This particular version of the PCPI protocol has been written for use in Cameroon. Another PCPI protocol has been submitted for Zambia with different sample sizes, but with the same approach.

Our aim with the PCPI studies is to evaluate a single-dose of malaria chemoprevention where genotypes (Pfdhps haplotypes ISGEAA and VAGKGS) are associated with SP resistance among healthy and symptom-free children between 3-5 years of age with unknown parasite status. In Cameroon, our objective is to measure parasite clearance and protection from infection conferred by malaria chemoprevention over a 63-day period in the presence/absence of the Pfdhps I431V mutation.

The new WHO chemoprevention guidelines remove the upper age limit of 12 months so that countries may evaluate PMC among a broader range of ages. We selected an age range for eligibility from 3 years and 0 days to 4 years and 364 days with the rationale being that 3-4 years old are more likely to tolerate PMC dosing better than children 0-2 years old. They are also more likely to have some modest level of semi-immunity and, therefore, are less likely to develop a clinical episode of malaria during the follow-up period relative to children who are 0-2 years of age.

After screening for eligibility, asymptomatic children based on a clinical examination and temperature reading will be randomised into one of four treatment groups on Day minus 7 (see Box 1). Children randomised to Groups 1-2 will receive placebo artesunate monotherapy for seven consecutive days. On Day 0, children in Groups 1-2 will then be given antimalarial chemoprevention therapy. In contrast, children randomised into Group 3 will receive active artesunate monotherapy for seven consecutive days and SP placebo on Day 0. Group 3 will establish one sub-set of children who are parasite-free at Day 0, and allow for an accurate estimate of background incidence (reflecting transmission intensity) to which all groups will be exposed during follow up. In addition, this group allows a more accurate estimation of underlying frequency of Pfdhps 431V mutations in the parasite population. Part of the rationale, as well, is to look at parasite clearance among those who were qPCR-positive at Day 0 and time to incident infection among qPCR-negative at Day 0. This will inform parameters of models we will use in data analysis. All children in Groups 1-3 will be followed 70 days total, 63 days (9-week period total) following treatment.

Box 1: Summary of treatments and children per group Group Treatment No. Children

1. sulfadoxine-pyrimethamine (SP)1 450
2. sulfadoxine-pyrimethamine plus amodiaquine (SPAQ)1 250
3. artesunate monotherapy (AS)2 200

Sample collection will be conducted at scheduled visits on Days 0, 2, 5, 7, 14, 21, and 28 visits as children provide a pin-prick of blood for a film slide and a dried blood-spot (DBS) on filter paper. On Days 35, 42, 49, 56, and 63 visits, only DBS will be collected. A study physician will be available 24 hours a day for unscheduled visits to review study subjects who develop symptoms.

All children will be screened for malaria symptoms, including a temperature check, at all contacts - scheduled visits and unscheduled visits - during their involvement in the study. All symptomatic children will have a malaria rapid diagnostic test (RDT) administered and a blood film taken. If a child is RDT-positive at any scheduled or unscheduled visit, the RDT will be stored for future genotyping rather than collecting a separate DBS. In all instances of a positive RDT, children will receive a full course of first-line therapy, artemether-lumefantrine (AL). Children who have an RDT diagnosis will no longer contribute to any future endpoints of the trial, but they will be asked to continue with symptom screening for the full follow-up period to Day 63 and, if symptomatic, they will be tested by RDT and again treated with first-line therapy if found positive and at least 28 days have elapsed since their previous AL-treated febrile episode. Where a child has a second febrile episode within 28 days with RDT-confirmed recurrent parasitaemia, the second-line treatment in Cameroon, artesunate-pyronaridine, will be administered. This ensures quality care is equitable for all participants, regardless of treatment group allocation.

The duration of follow-up in the PCPI protocol was carefully considered. Most study designs of malaria treatment efficacy have a primary endpoint of parasitaemia (present/absent) measured by slide microscopy at Day 28 (4 weeks) with PCR correction, an approach also outlined in the new WHO chemoprevention efficacy study (CPES) protocol.15 This study is consistent with procedures for the PCPI protocol. Consequently, data derived from PCPI studies will be comparable with data from other studies, including those conducted using the CPES protocol. The CPES protocol defines chemoprevention efficacy as both the ability to clear existing parasites and prevent a new infection for a short period (of 28 days). However, PCPI studies will separate resistance effects on these two outcomes of clearance and protection and extend the follow up period to Day 63 (9 weeks). This allows for better quantification of the protective efficacy against new infections by genotype, particularly when the mean duration of protection against more sensitive strains is higher or close to 28 days. Additionally, the choice of a 63-day follow-up simulates what might be the protective efficacy in a scenario where chemoprevention is administered to children every two months. This will be increasingly important for comparison purposes through meta-analysis as longer-acting interventions, including introduction of monoclonal therapies and malaria vaccines.

ELIGIBILITY:
Inclusion Criteria:

* Be 3-5 years old
* Exhibit no symptoms of malaria
* Have parents/guardians willing to have their child participate in all follow-up visits and seek care from study staff
* Reside in the study catchment area

Exclusion Criteria:

* Have evidence of acute illness as determined by clinical examination
* Exhibit symptoms of malaria (axillary fever ≥ 37.5 °C and / or history of fever in past 48 hours)
* Have known allergy to study medications
* Have received antimalarial treatment or azithromycin within 28 days prior to screening
* Be concomitantly receiving co-trimoxazole (trimethoprim-sulfamethoxazole)
* Be categorised as severely malnourished according to WHO child growth standards

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 902 (Actual)
Dates: Start 2024-06-10 (Actual); Primary Completion 2024-12-25 (Actual); Study Completion 2025-03-05 (Actual)

PRIMARY OUTCOMES:
Parasite clearance | 28 days (total follow up 63 days post SP dose)
  Time to clearance of parasite genotypes among SP recipients who were positive on Day 0 by qPCR (presence/absence of Pfdhps I431V) and measured to Day 63
Protection from infection | 28 days (total follow up 63 days post SP dose)
  (a) Mean duration of SP protection against parasite genotypes determined by Pfdhps gene sequence presence/absence of Pfdhps K540E among SP recipients who were parasite-free on Day 0 by qPCR (b) Mean duration of symptom-free status among SP recipients who were parasite free on Day 0 by qPCR, stratified by parasite Pfdhps genotype at time of febrile malaria episode

SECONDARY OUTCOMES:
Parasite clearance | 7 days (day 0 until day 7)
  Time to clearance of parasite genotypes among SPAQ recipients positive at Day 0 by qPCR (presence/absence of Pfdhps I431V) and measured to Day 63
Protection from infection | 35 days (day 0 until day 38)
  (a) Mean duration of SPAQ protection by qPCR (b) Mean duration of symptom-free status among SPAQ recipients
Therapeutic efficacy outcomes | 28 days (day 0 until day 28)
  For SP: (a)Acute clinical and parasitological response (ACPR) at Day 28 by presence/absence of Pfdhps I431V (b) ACPR at Day 28 by presence/absence of Pfdhps I431V + Pfdhps A581G For SPAQ: ACPR at Day 28

CONTACTS AND LOCATIONS:
Overall Officials: R Matthew Chico, MPH, PhD, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (1):
- Malantouen District Hospital Catchment Area, Magba, Cameroon

REFERENCES:
- [Background] World Health Organization. WHO guidelines for malaria, 3 June 2022: World Health Organization, 2022.
- [Background] Aponte JJ, Schellenberg D, Egan A, Breckenridge A, Carneiro I, Critchley J, Danquah I, Dodoo A, Kobbe R, Lell B, May J, Premji Z, Sanz S, Sevene E, Soulaymani-Becheikh R, Winstanley P, Adjei S, Anemana S, Chandramohan D, Issifou S, Mockenhaupt F, Owusu-Agyei S, Greenwood B, Grobusch MP, Kremsner PG, Macete E, Mshinda H, Newman RD, Slutsker L, Tanner M, Alonso P, Menendez C. Efficacy and safety of intermittent preventive treatment with sulfadoxine-pyrimethamine for malaria in African infants: a pooled analysis of six randomised, placebo-controlled trials. Lancet. 2009 Oct 31;374(9700):1533-42. doi: 10.1016/S0140-6736(09)61258-7. Epub 2009 Sep 16. PMID 19765816
- [Background] Schellenberg D, Menendez C, Kahigwa E, Aponte J, Vidal J, Tanner M, Mshinda H, Alonso P. Intermittent treatment for malaria and anaemia control at time of routine vaccinations in Tanzanian infants: a randomised, placebo-controlled trial. Lancet. 2001 May 12;357(9267):1471-7. doi: 10.1016/S0140-6736(00)04643-2. PMID 11377597
- [Background] Chandramohan D, Owusu-Agyei S, Carneiro I, Awine T, Amponsa-Achiano K, Mensah N, Jaffar S, Baiden R, Hodgson A, Binka F, Greenwood B. Cluster randomised trial of intermittent preventive treatment for malaria in infants in area of high, seasonal transmission in Ghana. BMJ. 2005 Oct 1;331(7519):727-33. doi: 10.1136/bmj.331.7519.727. PMID 16195288
- [Background] Macete E, Aide P, Aponte JJ, Sanz S, Mandomando I, Espasa M, Sigauque B, Dobano C, Mabunda S, DgeDge M, Alonso P, Menendez C. Intermittent preventive treatment for malaria control administered at the time of routine vaccinations in Mozambican infants: a randomized, placebo-controlled trial. J Infect Dis. 2006 Aug 1;194(3):276-85. doi: 10.1086/505431. Epub 2006 Jun 30. PMID 16826474
- [Background] Kobbe R, Kreuzberg C, Adjei S, Thompson B, Langefeld I, Thompson PA, Abruquah HH, Kreuels B, Ayim M, Busch W, Marks F, Amoah K, Opoku E, Meyer CG, Adjei O, May J. A randomized controlled trial of extended intermittent preventive antimalarial treatment in infants. Clin Infect Dis. 2007 Jul 1;45(1):16-25. doi: 10.1086/518575. Epub 2007 May 29. PMID 17554695
- [Background] Mockenhaupt FP, Reither K, Zanger P, Roepcke F, Danquah I, Saad E, Ziniel P, Dzisi SY, Frempong M, Agana-Nsiire P, Amoo-Sakyi F, Otchwemah R, Cramer JP, Anemana SD, Dietz E, Bienzle U. Intermittent preventive treatment in infants as a means of malaria control: a randomized, double-blind, placebo-controlled trial in northern Ghana. Antimicrob Agents Chemother. 2007 Sep;51(9):3273-81. doi: 10.1128/AAC.00513-07. Epub 2007 Jul 16. PMID 17638703
- [Background] Grobusch MP, Lell B, Schwarz NG, Gabor J, Dornemann J, Potschke M, Oyakhirome S, Kiessling GC, Necek M, Langin MU, Klein Klouwenberg P, Klopfer A, Naumann B, Altun H, Agnandji ST, Goesch J, Decker M, Salazar CL, Supan C, Kombila DU, Borchert L, Koster KB, Pongratz P, Adegnika AA, Glasenapp Iv, Issifou S, Kremsner PG. Intermittent preventive treatment against malaria in infants in Gabon--a randomized, double-blind, placebo-controlled trial. J Infect Dis. 2007 Dec 1;196(11):1595-602. doi: 10.1086/522160. Epub 2007 Oct 25. PMID 18008242
- [Background] Mayor A, Serra-Casas E, Sanz S, Aponte JJ, Macete E, Mandomando I, Puyol L, Berzosa P, Dobano C, Aide P, Sacarlal J, Benito A, Alonso P, Menendez C. Molecular markers of resistance to sulfadoxine-pyrimethamine during intermittent preventive treatment for malaria in Mozambican infants. J Infect Dis. 2008 Jun 15;197(12):1737-42. doi: 10.1086/588144. PMID 18419347
- [Background] Gupta H, Macete E, Bulo H, Salvador C, Warsame M, Carvalho E, Menard D, Ringwald P, Bassat Q, Enosse S, Mayor A. Drug-Resistant Polymorphisms and Copy Numbers in Plasmodium falciparum, Mozambique, 2015. Emerg Infect Dis. 2018 Jan;24(1):40-48. doi: 10.3201/eid2401.170864. PMID 29260689
- [Background] Gosling RD, Gesase S, Mosha JF, Carneiro I, Hashim R, Lemnge M, Mosha FW, Greenwood B, Chandramohan D. Protective efficacy and safety of three antimalarial regimens for intermittent preventive treatment for malaria in infants: a randomised, double-blind, placebo-controlled trial. Lancet. 2009 Oct 31;374(9700):1521-32. doi: 10.1016/S0140-6736(09)60997-1. Epub 2009 Sep 16. PMID 19765815
- [Background] Naidoo I, Roper C. Mapping 'partially resistant', 'fully resistant', and 'super resistant' malaria. Trends Parasitol. 2013 Oct;29(10):505-15. doi: 10.1016/j.pt.2013.08.002. Epub 2013 Sep 9. PMID 24028889
- [Background] Oguike MC, Falade CO, Shu E, Enato IG, Watila I, Baba ES, Bruce J, Webster J, Hamade P, Meek S, Chandramohan D, Sutherland CJ, Warhurst D, Roper C. Molecular determinants of sulfadoxine-pyrimethamine resistance in Plasmodium falciparum in Nigeria and the regional emergence of dhps 431V. Int J Parasitol Drugs Drug Resist. 2016 Dec;6(3):220-229. doi: 10.1016/j.ijpddr.2016.08.004. Epub 2016 Sep 29. PMID 27821281
- [Background] ACCESS-SMC Partnership. Effectiveness of seasonal malaria chemoprevention at scale in west and central Africa: an observational study. Lancet. 2020 Dec 5;396(10265):1829-1840. doi: 10.1016/S0140-6736(20)32227-3. PMID 33278936
- [Background] World Health Organisation. Malaria chemoprevention efficacy study protocol. Geneva: World Health Organisation, 2022.
- [Background] World Health Organization. WHO policy recommendation on intermittent preventive treatment during infancy with sulphadoxine-pyrimethamine (SP-IPTi) for plasmodium falciparum malaria control in Africa: World Health Organization, 2010.
- [Background] Esu EB, Oringanje C, Meremikwu MM. Intermittent preventive treatment for malaria in infants. Cochrane Database Syst Rev. 2021 Jul 17;7(7):CD011525. doi: 10.1002/14651858.CD011525.pub3. PMID 34273901
- [Background] Sutherland CJ, Fifer H, Pearce RJ, bin Reza F, Nicholas M, Haustein T, Njimgye-Tekumafor NE, Doherty JF, Gothard P, Polley SD, Chiodini PL. Novel pfdhps haplotypes among imported cases of Plasmodium falciparum malaria in the United Kingdom. Antimicrob Agents Chemother. 2009 Aug;53(8):3405-10. doi: 10.1128/AAC.00024-09. Epub 2009 May 11. PMID 19433569
- [Background] Beshir KB, Muwanguzi J, Nader J, Mansukhani R, Traore A, Gamougam K, Ceesay S, Bazie T, Kolie F, Lamine MM, Cairns M, Snell P, Scott S, Diallo A, Merle CS, NDiaye JL, Razafindralambo L, Moroso D, Ouedraogo JB, Zongo I, Kessely H, Doumagoum D, Bojang K, Ceesay S, Loua K, Maiga H, Dicko A, Sagara I, Laminou IM, Ogboi SJ, Eloike T, Milligan P, Sutherland CJ. Prevalence of Plasmodium falciparum haplotypes associated with resistance to sulfadoxine-pyrimethamine and amodiaquine before and after upscaling of seasonal malaria chemoprevention in seven African countries: a genomic surveillance study. Lancet Infect Dis. 2023 Mar;23(3):361-370. doi: 10.1016/S1473-3099(22)00593-X. Epub 2022 Oct 31. PMID 36328000
- [Background] Chijioke-Nwauche I, Oguike MC, Nwauche CA, Beshir KB, Sutherland CJ. Antimalarial drug resistance markers in human immunodeficiency virus (HIV)-positive and HIV-negative adults with asymptomatic malaria infections in Port Harcourt, Nigeria. Trans R Soc Trop Med Hyg. 2021 May 8;115(5):531-537. doi: 10.1093/trstmh/trab061. PMID 33823558
- [Background] Wang P, Sims PF, Hyde JE. A modified in vitro sulfadoxine susceptibility assay for Plasmodium falciparum suitable for investigating Fansidar resistance. Parasitology. 1997 Sep;115 ( Pt 3):223-30. doi: 10.1017/s0031182097001431. PMID 9300459
- [Background] Kimura I, Miyamoto J, Ohue-Kitano R, Watanabe K, Yamada T, Onuki M, Aoki R, Isobe Y, Kashihara D, Inoue D, Inaba A, Takamura Y, Taira S, Kumaki S, Watanabe M, Ito M, Nakagawa F, Irie J, Kakuta H, Shinohara M, Iwatsuki K, Tsujimoto G, Ohno H, Arita M, Itoh H, Hase K. Maternal gut microbiota in pregnancy influences offspring metabolic phenotype in mice. Science. 2020 Feb 28;367(6481):eaaw8429. doi: 10.1126/science.aaw8429. PMID 32108090
- [Background] Waltmann A, McQuade ETR, Chinkhumba J, Operario DJ, Mzembe E, Itoh M, Kayange M, Puerto-Meredith SM, Mathanga DP, Juliano JJ, Carroll I, Bartelt LA, Gutman JR, Meshnick SR. The positive effect of malaria IPTp-SP on birthweight is mediated by gestational weight gain but modifiable by maternal carriage of enteric pathogens. EBioMedicine. 2022 Mar;77:103871. doi: 10.1016/j.ebiom.2022.103871. Epub 2022 Feb 23. PMID 35217408
- [Background] Gimnig JE, MacArthur JR, M'bang'ombe M, Kramer MH, Chizani N, Stern RS, Mkandala C, Newman RD, Steketee RW, Campbell CH. Severe cutaneous reactions to sulfadoxine-pyrimethamine and trimethoprim-sulfamethoxazole in Blantyre District, Malawi. Am J Trop Med Hyg. 2006 May;74(5):738-43. PMID 16687672
- [Background] Taylor WR, White NJ. Antimalarial drug toxicity: a review. Drug Saf. 2004;27(1):25-61. doi: 10.2165/00002018-200427010-00003. PMID 14720085
- [Background] Adeleke OT, Oyenuga A, Slusher TM, Gbadero DA. Cluster-randomized controlled trial of intermittent preventive treatment in infancy using sulfadoxine-pyrimethamine (SP-IPTi): a pilot study in Nigeria. J Trop Pediatr. 2022 Dec 5;69(1):fmad001. doi: 10.1093/tropej/fmad001. PMID 36633492
- [Background] Wilson AL; IPTc Taskforce. A systematic review and meta-analysis of the efficacy and safety of intermittent preventive treatment of malaria in children (IPTc). PLoS One. 2011 Feb 14;6(2):e16976. doi: 10.1371/journal.pone.0016976. PMID 21340029
- [Background] Cairns M, Cisse B, Sokhna C, Cames C, Simondon K, Ba EH, Trape JF, Gaye O, Greenwood BM, Milligan PJ. Amodiaquine dosage and tolerability for intermittent preventive treatment to prevent malaria in children. Antimicrob Agents Chemother. 2010 Mar;54(3):1265-74. doi: 10.1128/AAC.01161-09. Epub 2010 Jan 11. PMID 20065053
- [Background] Bakai TA, Thomas A, Iwaz J, Atcha-Oubou T, Tchadjobo T, Khanafer N, Rabilloud M, Voirin N. Effectiveness of seasonal malaria chemoprevention in three regions of Togo: a population-based longitudinal study from 2013 to 2020. Malar J. 2022 Dec 31;21(1):400. doi: 10.1186/s12936-022-04434-w. PMID 36587191
- [Background] Sokhna C, Cisse B, Ba el H, Milligan P, Hallett R, Sutherland C, Gaye O, Boulanger D, Simondon K, Simondon F, Targett G, Lines J, Greenwood B, Trape JF. A trial of the efficacy, safety and impact on drug resistance of four drug regimens for seasonal intermittent preventive treatment for malaria in Senegalese children. PLoS One. 2008 Jan 23;3(1):e1471. doi: 10.1371/journal.pone.0001471. PMID 18213379
- [Derived] Martinez-Vega R, Mbacham WF, Ali I, Nji A, Mousa A, Beshir KB, Chopo-Pizarro A, Kaur H, Okell L, Hansson H, Hocke EF, Alifrangis M, Gosling R, Roper C, Sutherland C, Chico RM. Parasite clearance and protection from Plasmodium falciparum infection (PCPI): a three-arm, parallel, double-blinded, placebo-controlled, randomised trial of presumptive sulfadoxine-pyrimethamine versus sulfadoxine-pyrimethamine plus amodiaquine versus artesunate monotherapy among asymptomatic children 3-5 years of age in Cameroon. BMC Infect Dis. 2024 Sep 26;24(1):1028. doi: 10.1186/s12879-024-09868-y. PMID 39327613